CLINICAL TRIAL: NCT01762956
Title: Pelvic Floor Muscles Training in Men Undergoing Radiotherapy for Prostate Cancer: Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unobtainable sample size
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Aline Moreira Ribeiro, Physiotherapist, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 162/2015
Record Dates: First submitted 2013-01-03; First posted 2013-01-08 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer; Urologic Diseases
Keywords: Pelvic floor; Physical Therapy; Prostate cancer; Radiotherapy; Nuclear magnetic resonance
MeSH Terms: conditions — Prostatic Neoplasms; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (TG) (Experimental): The group of patients undergoing radiotherapy and submitted to pelvic floor muscles training.
  Interventions: Other: Pelvic floor muscles training
- Control group(CG) (No Intervention): The group of patients undergoing radiotherapy only.

INTERVENTIONS:
Other: Pelvic floor muscles training — The supervised muscle training will be conducted once a week with 45 minutes each session during the RT (12 weeks). In addition to the supervised sessions, patients will be instructed about the practice of home exercises and receive a guidance booklet of exercises with explanations of each exercise to be performed. These exercises must be performed daily and should be written down in the worksheet when they are performed. After this 3 month period, the patients will be encouraged to continue the exercise protocol at home without supervision. They must attend monthly to monitor adherence to home exercises.
  Arms: Training group (TG)

SUMMARY:
The pelvic floor disorders are a major problem in our current society with manifestations of micturition disorders, defecatory problems and sexual dysfunction. The pelvic floor muscles training arouses interest due the few studies on this subject. Studies are being conducted with emphasis on the post-prostatectomy urinary disorders, however, not associated with radiotherapy. The study of the effect of radiotherapy in these muscles is still uncertain. At right, we do not know if the effect of radiation can trigger important anatomical changes that could lead to pelvic floor disorders manifesting clinically as defecatory and urinary disorders. These issues motivate us to research, focusing on the evaluation of these muscles through magnetic nuclear resonance considering that radiation therapy has been increasingly used as a therapeutic option in the treatment of prostate cancer. The primary objective of this is to verify the effect of pelvic floor muscles training (PFMT) tract symptoms (LUTS), anorectal and sexual complaints in men with prostate cancer (PCa) treated with radiotherapy (RT). Secondly, the objective is to evaluate the effect of PFMT in its function and in the severity of urinary incontinence (UI) and evaluate the quality of life. The assessment of the changes occurred by the effect of radiation separately and jointly to the training of the pelvic floor muscles can help us to better understand some of the dysfunctions presented in this sample of patients as well as understanding the effect and the possible contribution of training of these muscles for treatment and/or prevention of these disorders.

DETAILED DESCRIPTION:
This present research is a randomized controlled clinical trial to be held in Clinics Hospital of Medical School of Ribeirão Preto - University of São Paulo (HCFMRP-USP) including men with confirmed diagnosis of prostate cancer by biopsy and having clinical indication for radiotherapy treatment (RT) who follow-up in the HCFMRP-USP and voluntarily consent to participate in this research. After consent, each patient must sign the consent term and then will be allocated by randomization in one of the following study groups:

* Training group (TG): the group of patients undergoing radiotherapy and submitted to pelvic floor muscles training;
* Control group (CG): the group of patients undergoing radiotherapy only. This research consists in four assessment: (1) Assessment 01: before started of radiotherapy; (2) Assessment 02: after two weeks started of RT; (3) Assessment 03: 03 months after started of RT (4) Assessment 04: 06 months after started of RT. All these assessments will be common for the participants of the research independently from the group they belong.

In each assessment, images of the pelvic floor muscles will be acquired by nuclear magnetic resonance. Parallel to the MRI, there will be a clinical assessment of the patient which consist of anamnesis and physical examination, where the assessment of pelvic floor muscle function will be tested objectively using a perineometer to evaluate the peak and the mean contraction as well as the duration of the performed sustained contraction. Data will be collected from three contractions, whose mean value will be used for this study. The myoelectric activity will be evaluated using electromyography biofeedback with electromyography anal probes. The patient will also answer a quality of life questionnaire (EORTC QLQ-C30 e PR25) and the others questionnaire: ICIQ-SF, QS-M and Jorge-Wexner Scale.

The patient of TG will be included in a supervised training protocol of the pelvic floor muscles. This protocol will be conducted in conjunction with the radiotherapy sessions.

The supervised muscle training will be conducted once a week with 45 minutes each session during the RT (12 weeks - 3 months). In addition to the supervised sessions, patients in this group will be instructed about the practice of home exercises and receive a guidance booklet of exercises with explanations of each exercise to be performed. These exercises must be performed daily and should be written down in the worksheet when they are performed. After this 3 month period, the patients will be encouraged to continue the exercise protocol at home without supervision. They must attend monthly to monitor adherence to home exercises.

The control group (CG) patients will not be instructed to perform pelvic floor exercises, instead they will only be assessed within the stipulated time.

ELIGIBILITY:
Inclusion Criteria:

* Men aged equal or higher than 45 years-old with confirmed diagnosis of prostate cancer by biopsy and having clinical indication for radiotherapy who follow-up in the HCFMRP-USP;
* No age distinction of race, creed and education;
* Men with graduation of PFM function greater than or equal to grade 2 evaluated by anal digital palpation (Oxford Scale Modified);
* Men who voluntarily consent to participate in research.

Exclusion Criteria:

* Men with anatomical abnormalities in perineal region due sequelae of surgery, pathology, trauma or injury sites;
* Men with associated neurological pathologies;
* Indication for adjuvant or rescue RT (radical prostatectomy);
* Men with acquired immune deficiency syndrome;
* PFMT carried out previously;
* Men with cardiac pacemakers, aneurysm clips, neurostimulators or other factors that preclude the application of review procedures established in this study;
* Men who have not completed proposed radiotherapy treatment;
* Men who do not accept to participate in this study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in the in the LUTS, anorectal and sexual complaints in six months. | 6 months after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Aline M Ribeiro, Principal Investigator — USP Ribeirão Preto; Harley F Oliveira, M.D., Study Director — USP Ribeirão Preto
Locations (1):
- Clinical Hospital of Medical College of Ribeirão Preto (HCFMRP), Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Bo K. Pelvic floor muscle strength and response to pelvic floor muscle training for stress urinary incontinence. Neurourol Urodyn. 2003;22(7):654-8. doi: 10.1002/nau.10153. PMID 14595609
- [Background] Centemero A, Rigatti L, Giraudo D, Lazzeri M, Lughezzani G, Zugna D, Montorsi F, Rigatti P, Guazzoni G. Preoperative pelvic floor muscle exercise for early continence after radical prostatectomy: a randomised controlled study. Eur Urol. 2010 Jun;57(6):1039-43. doi: 10.1016/j.eururo.2010.02.028. Epub 2010 Mar 1. PMID 20227168
- [Background] Dorey G, Glazener C, Buckley B, Cochran C, Moore K. Developing a pelvic floor muscle training regimen for use in a trial intervention. Physiotherapy. 2009 Sep;95(3):199-209. doi: 10.1016/j.physio.2009.03.003. Epub 2009 Jul 8. PMID 19635340
- [Background] Glazener C, Boachie C, Buckley B, Cochran C, Dorey G, Grant A, Hagen S, Kilonzo M, McDonald A, McPherson G, Moore K, Norrie J, Ramsay C, Vale L, N'Dow J. Urinary incontinence in men after formal one-to-one pelvic-floor muscle training following radical prostatectomy or transurethral resection of the prostate (MAPS): two parallel randomised controlled trials. Lancet. 2011 Jul 23;378(9788):328-37. doi: 10.1016/S0140-6736(11)60751-4. Epub 2011 Jul 7. PMID 21741700